CLINICAL TRIAL: NCT02095704
Title: Pharmacokinetics of a Standard Paracetamol Tablet and Oral Solution After Oral Administration in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Feifan Xie, Institute of Drug Metabolism and Pharmacokinetics,School of Pharmaceutical Sciences,Central South University, Central South University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CSU-YXY-001
Record Dates: First submitted 2014-03-19; First posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Focus of Study: Pharmacokinetics Analysis, in Vivo Dissolution Studies
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paracetamol oral solution (Experimental): dosage form: paracetamol oral solution;dosage:15.6ml(containing 500 mg of the active ingredient);frequency:single dose
  Interventions: Drug: paracetamol oral solution
- paracetamol tablet (Experimental): dosage form: paracetamol tablet;dosage: 500 mg;frequency:single dose
  Interventions: Drug: paracetamol tablet

INTERVENTIONS:
Drug: paracetamol oral solution — dosage form: paracetamol oral solution;dosage:15.6ml(containing 500 mg of the active ingredient);frequency:single dose
  Arms: paracetamol oral solution
Drug: paracetamol tablet — dosage form: paracetamol tablet;dosage: 500 mg;frequency:single dose
  Arms: paracetamol tablet

SUMMARY:
Drug dissolution in vivo play a crucial role for the bioavailability and therapeutic of an orally administered solid dosage form. The aim of this study was to evaluate the pharmacokinetics of a standard paracetamol tablet in comparison with oral solution in Chinese healthy volunteers. Based on the Noyes-Whitney equation and pharmacokinetics parameters, investigators trend to propose a method to estimate in vivo dissolution time and dissolution kinetics of solid dosage form.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: Male or female (limited to PK study)
2. Healthy volunteers, age: 18-45（medical history, physical examination, vital signs, ECG and lab tests are qualified during screening）
3. Body Mass Index（BMI）:19~24 or body weight is not less than 50Kg
4. Non-pregnant women confirmed by pregnancy test
5. Vital Signs: after 3 minutes supination, the following measurements criteria should be within ranges: body temperature (axillary temperature), 36.0~37.0 ℃; blood pressure, SBP 90~140mmHg（12.0~18.7kpa）and DBP 60~90mmHg（8.0~12.0kpa）; arterial pulse: 60~100 bpm
6. Non-hypersensitivity to this product or its similar product
7. Non-smoker, non-alcoholic
8. Subject must be able to sign Inform Consent prior to participation into this study
9. Subject must be able to communicate with investigator and comply with study protocol.

Exclusion Criteria:

Subjects meet with one or several of the following criteria should be excluded:

1. Subjects failed in physical examination
2. Pregnant or nursing women
3. Administration of a known drug that can cause damage to organs within 3 months
4. Administration of any prescription drug or non-prescription drug 2 weeks before initial dose
5. Before initial dose, participation in any other clinical trials within 3 months
6. Blood donation 3 months before this study, or plan to have blood donation during or one month after this study
7. Diagnosis of clinical evident diseases 2 weeks before initial dose
8. Primary diseases to vital organs
9. Physically or mentally disabled
10. Medical history of specific allergy (asthma, measles, eczematous dermatitis), or known to allergic to similar (including excipients)
11. Any other surgical or internal medicinal conditions that might cause damage to study subjects or will change the absorption, distribution, metabolism and elimination of investigational drug, including:

    * inflammatory intestinal syndrome, peptic ulcer, alimentary tract hemorrhage
    * a history of severe gastrointestinal tract operation, such as gastrectomy, gastrosmoty / jejunostomy or large bowel resection
    * a history of hepatic disease or laboratory examination findings such as ALT, AST, γ-GT or T-Bili showing clinically significant abnormalities to liver
    * a history of renal disease or laboratory examination findings such as creatinine, urea nitrogen, or albuminuria showing clinically significant abnormalities to kidney
    * urination disorder or dysuresia.
12. A history of immunological deficiency disease, or HIV positive
13. HBV or HCV positive
14. Women undergone menstrual period during study
15. Consumption of a significant amount of smoking or drinking, that is drinking more than 28 units of alcohol per week (1 unit: 285ml of beer, 25ml of liquor, or 1 glass of wine), or smoking more than 2 cigarettes
16. Frequent use of sedatives, hypnotics, stabilizers or other addictive drugs
17. Consumption of more than 8 cups of tea, coffee, and or caffeine beverages
18. Unable to complete this study for any others reasons.
19. Investigators.

Ages: 19 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
AUC | one month
  AUC:the area under the concentration-time curve
Cmax | one month
  Cmax: maximum plasma concentration
Tmax | one month
  Tmax: the time point of maximum plasma concentration
MRT | one month
  MRT: mean residence time